CLINICAL TRIAL: NCT06796621
Title: Effectiveness of Co-designed Anti-cyberbullying Intervention [Building Respectful Online Space (BROS)] Among Adolescents: A Feasibility Study
Brief Title: Building Respectful Online Space (BROS): Evaluating a Co-designed Anti-cyberbullying Intervention Among Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Concordia Lutheran School (Unknown)
Responsible Party: Principal Investigator, Lau Ying, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUHK-2025-YL
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cyberbullying
Keywords: Cyberbullying; Prevention; Adolescent
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Intervention Model Description: We will randomized two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Building Respectful Online Space (BROS) (Experimental): The intervention group participants will receive the BROS intervention across three sessions, depending on the school schedule, presented in a hybrid mode. The sessions focus on integrating psychoeducation, behavioural-specific cognitions, serious games, music, and reflection, as a means against cyberbullying. The content includes knowledge related to cyberbullying and online safety, cyberbullying coping skills, relationship skills, emotion management, and empathy towards victims through classroom sessions, short videos, serious games, and online musical therapy.
  Interventions: Behavioral: Building Respectful Online Space (BROS)
- Healthy diet education program (Placebo Comparator): For the control group participants, an alternative intervention (a healthy diet education program) with content unrelated to cyberbullying prevention will be given. The control group participants will receive the alternative intervention across three sessions. The content is based on recommendations from the Centre for Health Protection, the Government of the Hong Kong Special Administrative Region (CHP, 2024) on healthy eating pyramids, emotional eating, healthy weight management, and nutritional requirements for adolescents.
  Interventions: Behavioral: Healthy diet education program

INTERVENTIONS:
Behavioral: Building Respectful Online Space (BROS) — Session 1 (40 minutes to 50 minutes): Respectful online relationship (Psychoeducation) using face-to-face approach with 40 minutes to 50 minutes online serious game Session 2 (40 minutes to 50 minutes): Navigating the online world (Psychoeducation) using face-to-face approach with 20 to 30 minutes online music therapy Session 3 (40 minutes to 50 minutes): Behaviour specific cognitions and reflection using face-to-face approach
  Arms: Building Respectful Online Space (BROS)
Behavioral: Healthy diet education program — Session 1 (40 - 50 minutes): Healthy Diet Pyramid (Psychoeducation) using face-to-face approach Session 2 (40 - 50 minutes): Mindful Eating and Healthy Weight Management (Psychoeducation) using face-to-face approach Session 3 (40 - 50 minutes): Healthy Eating Habits for Life (Psychoeducation)using face-to-face approach
  Arms: Healthy diet education program

SUMMARY:
Background: The growing prevalence of cyberbullying throughout the world indicates the importance of anti-cyberbullying interventions, especially for adolescents. While few interventions target cyberbullying, content from different regions may not necessarily apply to local contexts, adolescents' viewpoints were not considered in the past designs, few local RCTs, and unclear sustainability.

Objectives: To evaluate the feasibility, acceptability and preliminarily effects of the co-designed anti-cyberbullying intervention: Building Respectful Online Space (BROS).

Methods: A sample of around 90 aged 12 to 15 will be recruited from secondary schools in Hong Kong. This study will adopt a 2-arm experimental trial. Each class will be randomly assigned equally into the intervention arm (BROS) and control arm (Heathy Diet), and eligible students will be allocated to either arm accordingly. The intervention will be provided in one or 3 days based on the school schedule. Participants will be assessed at baseline, 3 weeks later, and 12-week follow-up assessments. The primary outcome is cyberbullying behaviour of perpetration and victimisation; the secondary outcome includes cyberbullying attitudes, sleep quality, and psychosocial well-being. Feasibility and acceptability will be assessed. And generalised estimating equations analysis will be used to investigate the research objectives.

Potential contributions: The results of this study will provide evidence-based support for using a blended approach to prevent cyberbullying, promote psychosocial well-being, and promote sleep health. This intervention is dedicated to using evidence-to-user-driven ideas to develop culturally sensitive interventions to effectively prevent cyberbullying in the future.

DETAILED DESCRIPTION:
There is a growing body of literature that recognises whole-school strategy can be effective in preventing cyberbullying. Interventions, such as NoTrap! in Italy, Prev@cib in Spain, Media Heroes in Germany, 'Friendly Attac' in Belgium , and ViSC in Austria, have been shown to effectively prevent cyberbullying. Some school-based programmes integrate digital format into their intervention; for instance, the 'Cyber Friendly Schools' intervention in Australia utilises the online modules to facilitate learning; the 'Friendly Attac' program incorporates series games, and a study adopted a purely online approach to prevent cyberbullying in the Netherlands. A recent systematic review suggests that school-based intervention could comprehensively promote healthy online behaviours and reduce cyberbullying incidence among adolescents .

ELIGIBILITY:
Inclusion Criteria:

* Students in 1st to 3rd grades in secondary schools
* Students are able to read and understand Chinese
* Students obtained informed consent signed by their parents or legal guardians

Exclusion Criteria:

* Students in grades 4th through 6th who are heavily involved in homework and examination
* Students with severe diseases or co-occurring disorders
* Students' parents/ legal guardians who refuse to sign informed consent.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cyberbullying behaviour | Baseline, pre-intervention, immediately after the intervention, and 3 months follow-up assessment after intervention
  The Cyberbullying Behaviour Scale (CBBS) consists of E-Victimisation Scale (E-VS) and the E-Bullying Scale (E-BS), is the validated 11-item scale for measuring cyberbullying behaviour. The scale consist of two domain: 5-item of E-VS and 6-item of E-BS for adolescents with a 7-point Likert scale (Lam & Li, 2013) that measure cyberbullying victimization and perpetration respectively. The sum score for E-VS range from 5-35, and E-BS from 5-42, and a higher score indicate severity of respective cyberbullying behavior (Lam & Li, 2013). The Chinese version of CBBS will be used that was translated and validated by our research team.

SECONDARY OUTCOMES:
Cyberbullying attitude | Baseline, pre-intervention, immediately after the intervention, and 3 months follow-up assessment after intervention
  Cyberbullying Attitude Scale (CBAS) is used to identify positive cyberbullying attitude. The CBAS is a 9-item self-report scale using a 5-point Likert scale (Barlett et al., 2016). It consists of 5 items for harmful cyberbullying attitudes (HCA), which assess individuals' perceptions of cyberbullying perpetration, and 4 items for general cyberbullying characteristics (GCC). The range of HCA scores from 5 to 25 and the range of GCC scores from 4 to 20. A higher score indicates more harmful cyberbullying attitudes. The Chinese version of CBAS will be used that was translated and validated by our research team.
Sleep outcomes: Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction | Baseline, pre-intervention, immediately after the intervention, and 3 months follow-up assessment after intervention
  The Chinese version of Pittsburgh Sleep Quality Index (PSQI) will be used to assess subjective sleep disruption and quality throughout the previous month (Ho et al., 2021). Subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disruptions, sleep medication, and daytime dysfunction are the seven components that comprise the components of the PSQI. The range of scores for each item is 0 (no difficulty) to 3 (extreme difficulty). The total score ranges between 0 and 21. Poorer quality of sleep is indicated by a higher overall score.
Mental well-being | Baseline, pre-intervention, immediately after the intervention, and 3 months follow-up assessment after intervention
  The Chinese version of the WHO 5-item Well-Being Index is used to assess participants' mental well-being (Fung et al., 2022). Each item is rated on a six-point Likert scale, ranging from 0 (at no time) to 5 (always), the total score range from 0 to 25. A higher score indicates greater mental well-being.
Life satisfaction | Baseline, pre-intervention, immediately after the intervention, and 3 months follow-up assessment after intervention
  The Chinese version of the Satisfaction With Life Scale (SWLS) (SWLS) is used to assess global cognitive judgments of satisfaction with one's life (Sachs, 2003).It consists of 5 items with a 7-item Likert scale (Pavot & Diener, 1993), ranging from 1 (strongly disagree) to 7 (strongly agree) . The total score ranges from 7 to 35, with a higher score represent grater social well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Given that it is a very preliminary stage, the authors undecided to share IPD at this stage.